CLINICAL TRIAL: NCT06618651
Title: Phase I Study of Safety, Tolerability, Pharmacokinetics and Efficacy of SHR-3821 Injection in Subjects With Advanced Solid Tumors
Brief Title: A Study of SHR-3821 Injection in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-3821-101
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: To evaluate the safety, tolerability, pharmacokinetics and efficacy of SHR-3821 injection in subjects with advanced solid tumors.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-3821 injection (Experimental)
  Interventions: Drug: SHR-3821 injection

INTERVENTIONS:
Drug: SHR-3821 injection — SHR-3821 injection

SUMMARY:
This is an open label, multi-center, multiple dose Phase I study to evaluate the safety, tolerability, pharmacokinetics and efficacy of SHR-3821 injection in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and written informed consent.
2. 18-75 years older, no gender limitation.
3. Eastern Cooperative Oncology Group (ECOG) score: 0-1.
4. With a life expectancy ≥ 3 months.
5. Pathologically diagnosed advanced solid tumor.
6. Be able to provide fresh or archived tumour tissue.
7. At least one measurable lesion according to RECIST v1.1.
8. Adequate bone marrow reserve and organ function.
9. Contraception is required during the trial.

Exclusion Criteria:

1. Meningeal metastasis history or clinical symptoms of central nervous system metastasis.
2. Uncontrollable tumor-related pain.
3. Uncontrolled pleural effusion, pericardial effusion, or abdominal effusion with clinical symptoms.
4. Received systemic antitumor therapy before the first dose.
5. Treated with similar target therapy as SHR-3821 before the first dose.
6. Received systemic anticancer treatments 4 weeks prior to the initiation of the study treatment.
7. Unresolved CTCAE 5.0>=grade 2 toxicities from previous anticancer therapy.
8. Current or History of ILD.
9. Active severe digestive disease.
10. Previous or co-existing malignancies.
11. History of severe hypersensitivity reactions to either the drug substances or inactive ingredients of SHR-3821.
12. Active hepatitis B or active hepatitis C.
13. Other inappropriate situation considered by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
DLT | 3 weeks
AE | Screening up to study completion, an average of 1 year
MTD | 3 weeks
RP2D | Screening up to study completion, an average of 1 year

SECONDARY OUTCOMES:
Blood concentration of SHR-3821 after single and continuous administration | Screening up to study completion, an average of 1 year
PK parameters of SHR-3821 after single and continuous administration: Tmax | Screening up to study completion, an average of 1 year
PK parameters of SHR-3821 after single and continuous administration: Cmax | Screening up to study completion, an average of 1 year
PK parameters of SHR-3821 after single and continuous administration: AUC0-t | Screening up to study completion, an average of 1 year
Drug Resistant Antibody (ADA) to SHR-3821 | Screening up to study completion, an average of 1 year
Objective response rate (ORR) | Screening up to study completion, an average of 1 year
Disease control rate (DCR) | Screening up to study completion, an average of 1 year
Progression-free survival (PFS) | Screening up to study completion, an average of 1 year
Overall survival (OS) | Screening up to study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided